CLINICAL TRIAL: NCT05471466
Title: Scar Outcomes for Scalpel Versus Diathermy Neck Incisions in an Afro-Caribbean Population: A Randomized Controlled Trial
Brief Title: Scar Outcomes for Scalpel Versus Diathermy Neck Incisions in an Afro-Caribbean Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CeLois Lawrence (Other)
Collaborators: The University of The West Indies (Other)
Responsible Party: Sponsor-Investigator, CeLois Lawrence, Senior Resident- Department of Ear, Nose and Throat, Kingston Public Hospital
Organization: Kingston Public Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1
Record Dates: First submitted 2022-07-14; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Surgical Incision
Keywords: Skin Wound; Afro-Caribbean or black skin; Diathermy or electrosurgical unit; Neck surgery; Scalpel Wound
MeSH Terms: conditions — Surgical Wound; Fever

STUDY DESIGN:
Intervention Model Description: Randomized controlled double-blinded
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the participants nor the outcomes assessor were aware of which side of the incision was made using the scalpel or the electrosurgical unit device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diathermy- Electrosurgical Unit Cutting Settings (Active Comparator): One half of the neck incision in each participant was made using diathermy (electrosurgical unit cutting settings at 15 watts Blend One mode).
  Interventions: Procedure: Surgical incision
- Scalpel- Surgical Blade (Active Comparator): One half of the neck incision in each participant was made using a scalpel (size 10 surgical blade).
  Interventions: Procedure: Surgical incision

INTERVENTIONS:
Procedure: Surgical incision — Surgical incisions to the neck as part of the management of the head and neck condition.

SUMMARY:
This is randomized controlled double-blinded trial comparing the scar outcomes of diathermy versus scalpel surgical incisions in the neck. It was conducted in humans in an Afro-Caribbean (black) population.

DETAILED DESCRIPTION:
This double-blinded parallel group randomized controlled trial included consecutive eligible Ear, Nose and Throat (ENT) patients at a Jamaican tertiary hospital requiring an anterior neck incision. The purpose was to determine whether cutting diathermy adversely affected scar cosmesis in an Afro-Caribbean population and whether complexion influenced this outcome. Half of the incision in each of 35 patients was randomly assigned to either cutting electrocautery or scalpel. The patients and the assessor of the scars were blinded and the both sides of the scar were assessed by both parties using the patient component of the Patient and Observer Scar Assessment Score (PSAS) and the Vancouver Scar Scale (VSS) at 1 week, 3 months and 6 months postoperative intervals. The Fitzpatrick Phototyping Scale was used for skin pigmentation classification.

ELIGIBILITY:
Inclusion Criteria:

* The following are the conditions for inclusion in the study:

  1. Subjects must be 18 years of age or older and give written informed consent
  2. Treatment for surgical condition requires the type of neck incision that would be used for a standard thyroidectomy i.e. a horizontal incision about 2 fingers' breadth above the sternal notch or in a skin crease close to that landmark extending from the anterior border of one sternocleidomastoid muscle to another.
  3. Only elective surgical cases will be included
  4. Only primary incisions will be included i.e. no completion thyroidectomies or scar revisions to the neck
  5. Only clean surgeries will be included
  6. All wounds must be closed primarily i.e. no wounds healed by secondary intention or delayed primary closure or flap or graft coverage will be included

Exclusion Criteria:

* The following are conditions for exclusion from the study:

  1. Subjects with skin pathologies i.e. patients with dermatological conditions, skin infections, altered pigmentation to the neck, use of skin-lightening agents to the neck, or neurofibromatosis will be excluded.
  2. Surgeries requiring a drain (This is a relative exclusion criterion as subjects with drains that are pulled through skin outside of the incision site may be included. However, patient must consent to this prior).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Difference between diathermy and scalpel scar cosmesis- Total PSAS. | Six months
  Difference in scar cosmesis between the diathermy and scalpel sides of the scar as assesses by the Total Patient Scar Assessment Score (PSAS) on a scale of 6 to 60 where 6 is as per normal skin and 60 is very different from normal skin. There were measured at 1 week, 3 months, and 6 months post-surgery.
Difference between diathermy and scalpel scar cosmesis- Overall PSAS. | Six months
  Difference in scar cosmesis between the diathermy and scalpel sides of the scar as assesses by the Overall Patient Scar Assessment Score (PSAS) on a scale of 1 to 10 where 1 is as per normal skin and 10 is very different from normal skin. These were measured at 1 week, 3 months, and 6 months post-surgery.
Difference between diathermy and scalpel scar cosmesis- VSS. | Six months
  Difference in scar cosmesis between the diathermy and scalpel sides of the scar as assesses by the Vancouver Scar Scale (VSS) on a scale of 0 to 13 where 0 is as per normal skin and 13 is the most extreme difference from normal skin. These were measured at 1 week, 3 months, and 6 months post-surgery.

SECONDARY OUTCOMES:
Difference in scar cosmesis based on skin complexion. | Six months
  Difference in scar cosmesis based on Fitzpatrick Phototyping category (skin complexion) on a scale of 1 to 6 where 1 is the lightest skin complexion and 6 is the darkest. This is as per the Total Patient Scar Assessment Score (PSAS), Overall PSAS and the Vancouver Scar Scale (VSS) measured at 1 week, 3 months, and 6 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: CeLois Lawrence, BSc MBBS, Principal Investigator — Kingston Public Hospital
Locations (1):
- Kingston Public Hospital, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data directly related to the research outcomes in the publication will be shared upon request.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available up to 2 years after the date of publication/ journal issue.